CLINICAL TRIAL: NCT01352559
Title: Prediction of Antidepressant Response Using Pharmacogenetics of Bioamine Transporter and Peripheral Lymphocytic Phenotype
Brief Title: Prediction of Antidepressant Response Using Pharmacogenetics and Peripheral Lymphocytic Phenotype
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Doh Kwan Kim, M.D., pHD, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001-11-03
Record Dates: First submitted 2011-04-21; First posted 2011-05-12 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Depression
Keywords: Pharmacogenomics; Prediction of Antidepressant Response; Depressed Patients; biomarkers; phenotype; Antidepressant Response; Adverse Reaction to Drug
MeSH Terms: conditions — Depression; Drug-Related Side Effects and Adverse Reactions | interventions — Paroxetine; Milnacipran; Nortriptyline; Mirtazapine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- responders (Experimental): 50 ≤ Decrease rate(%) of HAM-D score
  Interventions: Drug: responders
- non-responders (Active Comparator): nonresponders is a patients having 50 > Decrease rate(%) of HAM-D score
  Interventions: Drug: non-responders

INTERVENTIONS:
Drug: responders — Antidepressants administration for 6 weeks under therapeutic dose
  Other Names: fluoxetine_Prozac; paroxetine_Paxil, Seroxat; sertraline_Zoloft; milnacipran; venlafaxine_Effexor; nortriptyline_Aventyl, Pamelor, Noritren; mirtazapine_Avanza, Zispin, Remeron
  Arms: responders
Drug: non-responders — Antidepressants administration for 6 weeks under therapeutic dose
  Other Names: SSRI nonresponders
  Arms: non-responders

SUMMARY:
The purpose of this study is to determine whether pharmacogenomic study of bioamine transporters and peripheral lymphatic biomarkers(phenotype) predict antidepressant responsiveness in advance before the appearance of the drug effects until 4~6 weeks after drug administration.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether genomic effects or peripheral lymphatic biomarkers on antidepressant response differed by class of drug, whether genomic and biomarker differences between drug responders and nonresponders predict the response of antidepressant and to construct the prediction model for antidepressant treatment in order to aid to select the their genetically or endophenotypic matching drugs.

ELIGIBILITY:
Inclusion Criteria:

1. eligible patients were enrolled in the clinical trials program of hte Samsung Medical Center Geropsychiatry and Affective Disorder Clinics(Seoul, Korea). They received a semistructured diagnostic interview, the Samsung Psychiatric Evaluation Schedule. The affective disorder section of the Samsung Psychiatric Evaluation Schedule uses the Korean version of the structured clinical interview for the diagnostic and statistical manual of mental disorders, Fourth edition.
2. interview with one more patient's family member for objective diagnosis and final diagnosis decision by agreements of two more psychiatric physicians

Exclusion Criteria:

1. received psychotropic medication within 2 weeks of the study or fluoxetine within 4 weeks
2. potential study participants for pregnancy, significant medical conditions, abnormal laboratory baseline values, unstable psychiatric features(eg.suicidal), history of alcohol of drug dependence, seizures, head trauma with loss of consciousness, neurological illness, or concomitant Axis I psychiatric disorder.

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2001-11; Primary Completion 2007-03 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Antidepressant Response at 6 weeks | 6 weeks
  antidepressant response is defined as the decrease rate of HAM-D score for 6week was = or > 50%
  Measurement Unit = responders, nonresponders

SECONDARY OUTCOMES:
Biological value at 0 and 6 weeks | 6 weeks
  Biological value is defined as
  1. Genetic information of bioamine transporter genes of patients. Measurement unit = if it is SNP,it is A, T, G, or C, and if VNTR, short or long allele
     or
  2. Biological measure value of patients at 0 and 6week after antidepressant treatment(ex. peripheral markers such as serum BDNF, CREB...).
  Measurement unit = numerical value and thier unit such as O.D.(Optical Density)

CONTACTS AND LOCATIONS:
Overall Officials: Doh Kwan Kim, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Kangnam, Seoul, South Korea